CLINICAL TRIAL: NCT00903253
Title: A Double-Blind, Placebo Controlled, Single, Escalating Dose Study to Evaluate the Preliminary Pharmacokinetics, Safety and Tolerability of LNK-754 in Healthy Elderly Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Link Medicine Corporation (Industry)
Allocation: Randomized | Masking: Double
Other Study IDs: LNK754-0901-1A
Record Dates: First submitted 2009-05-14; First posted 2009-05-18 (Estimated); Last update posted 2009-09-10 (Estimated); Status verified 2009-09

CONDITIONS: Healthy Elderly Volunteers
MeSH Terms: interventions — LNK-754

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: LNK-754

SUMMARY:
The objective of this study is to evaluate the single-dose plasma pharmacokinetics of LNK-754 as well as safety and tolerability in normal healthy male and female elderly volunteers

ELIGIBILITY:
Inclusion Criteria:

* Males and Females aged 60 to 75 years
* Good general health as determined by medical history and physical examination
* Body Mass Index of 18-32, inclusive
* Estimate of creatinine clearance by Cockcroft-Gault that is normal for age and sex (greater than or equal to 60mL/min)
* Normal hemoccult test at screening and baseline
* Voluntarily consent to participate in the study
* Willing to adhere to the protocol requirements

Exclusion Criteria:

* Subjects with clinically significant cardiovascular, pulmonary, renal, hepatic, gastrointestinal, neurological, sleep disorders by DSM-IV criteria, endocrine, hematological, or metabolic disease as determined by medical history and physical examination
* Subjects who have been diagnosed with or meet the Diagnostic and Statistical Manual of Mental Disorders Fourth Edition, Text Revision (DSM-IV_TR) criteria for any significant psychiatric or psychoactive substance use disorder within the past year
* Subjects with positive urine drug screen or compounds associated with abuse in the absence of medical justification for their presence
* QTcB greater than 450 msec (males), or greater than 470 (females), based on the average interval of triplicate ECGs obtained after five minutes rest in a supine position using hte ECG algorithm
* Clinically significant abnormal screening results or laboratory tests
* Pregnant or nursing or planning a pregnancy, or planning on fathering a child

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-05; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Plasma Pharmacokinetics | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- CEDRA Clinical Research, Austin, Texas, United States